CLINICAL TRIAL: NCT03741673
Title: A Phase III Trial of Pre-Operative Stereotactic Radiosurgery (SRS) Versus Post-Operative SRS for Brain Metastases
Brief Title: Pre-operative SRS or Post-operative SRS in Treating Cancer Patients With Brain Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0552; NCI-2018-02220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0552 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-11-09; First posted 2018-11-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Malignant Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Neoplasms; Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (pre-operative SRS) (Experimental): Patients undergo SRS within 30 days of randomization followed by surgery within 30 days. Patients may undergo additional SRS if disease returns after treatment.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery
- Group II (post-operative SRS) (Active Comparator): Patients undergo surgery within 30 days of randomization followed by standard of care SRS within 30 days. Patients may undergo additional SRS if disease returns after treatment.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This phase III trial studies stereotactic radiosurgery (SRS) before surgery to see how well it works compared with SRS after surgery in treating patients with cancer that has spread to the brain (brain metastases). SRS is the delivery of focused, high-dose radiation given in a single session to the tumors, with a minimal dose given to uninvolved areas of the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the 1 year leptomeningeal disease (LMD)-free rate among patients with surgically resectable metastatic brain lesions randomized to post-operative stereotactic radiosurgery (SRS) (standard care) versus pre-operative SRS followed by surgery (experimental arm).

SECONDARY OBJECTIVE:

I. To investigate the local control (LC), distant brain metastasis rate, overall survival (OS) of pre-operative (pre-op) versus (vs) post-operative (post-op) SRS in patients with brain metastasis.

EXPLORATORY OBJECTIVES:

I. To assess the reliability of different imaging features by using a combination of patient data and phantom data to quantify the uncertainties associated with using magnetic resonance imaging (MRI) for radiomics studies.

II. To assess the correlation of imaging-pathology correlates using multiparametric imaging that characterize the tumor and peri-tumoral microenvironment including features such as tumor vascular characteristics, cellular density, oxygenation and presence of inflammation/immune reactivity.

III. To investigate the neuro-cognitive impact, patient reported outcomes and health-related quality of life of pre-operative (pre-op) vs post-operative (post-op) SRS in patients with brain metastasis.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I (PRE-OPERATIVE SRS): Patients undergo SRS within 15 days of randomization followed by surgery within 15 days. Patients may undergo additional SRS if disease returns after treatment.

GROUP II (POST-OPERATIVE SRS): Patients undergo surgery within 15 days of randomization followed by standard of care SRS within 30 days. Patients may undergo additional SRS if disease returns after treatment.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* The primary lesion pre-operatively can have a maximum diameter of =< 4 cm for single fraction and =< 7 cm for multifraction therapy
* Patients must be considered candidates for SRS within +/- 30 days of surgical resection as defined by either history and physical (H&P) or presentation at brain metastasis tumor board conference note
* Patients must have a Karnofsky performance scores >= 70 or Eastern Cooperative Oncology Group (ECOG) >= 2 within 30 days of enrollment
* Patients must agree to randomization as documented by signing the Institutional Review Board (IRB) approved consent form
* No radiographic evidence of leptomeningeal disease on MD Anderson Cancer Center (MDACC) departmental radiology report or study neuro-radiologist review
* Documented history of malignancy

Exclusion Criteria:

* Patients who have received prior radiation therapy to the brain for any reason
* The primary tumor is small-cell lung cancer, lymphoma, leukemia, or multiple myeloma
* For females, if they are pregnant or breast-feeding (The exclusion is made because gadolinium may be teratogenic in pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Leptomeningeal disease (LMD)-free rate | At 1 year
  Aalen-Johansen estimates will be used for LMD. Uni- and multi-variable analysis of time to LMD will be done using Fine-Gray proportional hazards regression. Model assumptions will be verified graphically by residual analyses.

SECONDARY OUTCOMES:
Local control rate | At 1 year
  Aalen-Johansen estimates will be used for local recurrence. Uni- and multi-variable analysis of time to local recurrence will be done using Fine-Gray proportional hazards regression. Model assumptions will be verified graphically by residual analyses.
Distant brain control | At 1 year
  Aalen-Johansen estimates will be used for distant brain recurrence. Uni- and multi-variable analysis of time to distant brain recurrence will be done using Fine-Gray proportional hazards regression. Model assumptions will be verified graphically by residual analyses.
Overall survival (OS) | At 1 year
  Kaplan-Meier estimates will be utilized for survival. Uni- and multi-variable analysis of overall survival will be done with Cox proportional hazards regression.

OTHER OUTCOMES:
Delta radiomics | Up to 4 years
  Radiomic texture features and changes in features at diagnosis with pathology and over time will be included in various classifiers for modeling including decision trees, discriminate analysis, and nearest neighbor classifiers using classification learner in Matlab.
Circulating tumor cell analysis | Up to 4 years
Cerebral spinal fluid analysis | Up to 4 years
Neurocognitive function measured by HVLT-R questionnaire | Up to 1 year from start of treatment
  Measured by neurocognitive decline on Hopkins Verbal Learning Test-Revised (HVLT-R)
Symptom burden questionnaire | Up to 1 year from start of treatment
  Measured by the MD Anderson Symptom Inventory Brain Tumor (MDASI-BT).
Health outcomes questionnaire | Up to 1 year from start of treatment
  Measured by the European Quality of Life Five Dimension Five Level Scale questionnaire (EQ-5D-5L).
Neurocognitive function measured by COWA questionnaire | Up to 1 year from start of treatment
  Measured by neurocognitive decline on Controlled Oral Word Association (COWA)
Neurocognitive function measured by TMT questionnaire | Up to 1 year from start of treatment
  Measured by neurocognitive decline on and Trail Making Test (TMT) parts A and B
Neurocognitive function measured by CTB COMP questionnaire | Up to 1 year from start of treatment
  Measured by neurocognitive decline on Clinical Trial Battery Composite (CTB COMP) score.

CONTACTS AND LOCATIONS:
Overall Officials: Debra N Yeboa, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Yeboa DN, Li J, Lin R, Prabhu SS, Beckham TH, Woodhouse K, Swanson TA, Weinberg JS, Wang X, Chi X, Ejezie CL, Suki D, Wang C, Ene C, McCutcheon IE, McGovern S, McAleer MF, Tom M, Ghia A, Perni S, Jiang W, De B, Chung C, Kim BYS, O'Brien BJ, Huse JT, Wefel JS, Court L, Tawbi H, Janku F, Guha-Thakurta N, Debnam JM, Johnson J, Taslicay CA, Alvarez-Breckenridge C, Raza SM, Heimberger AB, DeMonte F, North R, Briere TM, de Groot JF, Sawaya R, Grosshans D, Lang FF, Rao G, Ferguson SD. Therapy, Safety, and Logistics of Preoperative vs Postoperative Stereotactic Radiation Therapy: A Preliminary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2025 Aug 1;11(8):890-899. doi: 10.1001/jamaoncol.2025.1770. PMID 40531511
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03741673/ICF_000.pdf